CLINICAL TRIAL: NCT06850831
Title: Effect of Intracoronary N-Acetylcysteine on Malondialdehyde, Interleukin-6, High Sensitivity Troponin I, Caspase-3, Global Longitudinal Strain, and 6-Minutes Walking Test in Patients With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: Effect of Intracoronary N-Acetylcysteine in Patients With ST-Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: dr. Ahmad Yasa, Sp.JP, Subsp.K.I.(K), M.Kes, FIHA, FasCC, FA (Other)
Responsible Party: Sponsor-Investigator, dr. Ahmad Yasa, Sp.JP, Subsp.K.I.(K), M.Kes, FIHA, FasCC, FA, Principal Investigator, Universitas Sebelas Maret
Organization: Universitas Sebelas Maret (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 374/II/HREC/2025
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: STEMI - ST Elevation Myocardial Infarction (MI); Primary PCI - STEMI
Keywords: STEMI; Primary PCI; Intracoronary NAC; Reperfusion Injury; Apoptosis; Necrosis; Oxidative Stress; Remodelling; Left ventricular dysfunction; Physical Recovery
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Reperfusion Injury; Necrosis; Ventricular Dysfunction, Left

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial and Double Blind (Researcher & Patients)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracoronary NAC (Experimental): The intervention group will have intracoronary NAC 480 mg immediately after the lesion is opened during primary PCI is performed besides standard treatment of STEMI before further evaluation.
- Control (Placebo Comparator): The intervention group will have intracoronary N-AC 480 mg immediately after the lesion is opened during primary PCI besides standard treatment of STEMI before further evaluation.
  Interventions: Drug: Antipac

INTERVENTIONS:
Drug: Antipac — The first group is the NAC group, which will get intracoronary NAC 480 mg immediately after the lesion is opened during primary PCI. And the second group will have placebo immediately after the lesion is opened during primary PCI.
  Arms: Control

SUMMARY:
Primary percutaneous coronary intervention (PCI) is the gold standard for reperfusion therapy in patients with ST-elevation myocardial infarction (STEMI), as it restores blood flow by clearing the blocked coronary artery. This process helps reoxygenate the previously hypoxic myocardium, potentially preventing further myocardial cell death. However, despite its benefits, reperfusion therapy, including primary PCI, can also lead to reperfusion injury, which may worsen myocardial damage, increase infarct size, and negatively impact patient outcomes. One of the key contributors to reperfusion injury is reactive oxygen species (ROS), which can induce oncosis, necrosis, and apoptosis, ultimately promoting cell death, myocardial remodeling, left ventricular systolic dysfunction and poorer clinical outcomes. N-Acetylcysteine (NAC), widely known for its mucolytic properties, has also been recognized for its antioxidant and cardioprotective effects. By reducing oxidative stress, NAC has been shown to decrease oncosis, necrosis, and apoptosis, as evidenced by lower levels of malondialdehyde, IL-6, troponin, caspase-3, and major adverse cardiac events in STEMI patients. However, existing research on NAC has only explored oral and intravenous administration. Given that reperfusion injury occurs rapidly, an optimal approach would involve delivering cardioprotective agents directly to the target site, specifically coronary artery endothelial cells. To date, no studies have directly investigated the effects of intracoronary NAC administration in STEMI patients undergoing primary PCI.

DETAILED DESCRIPTION:
This study is a double-blind, randomized controlled trial, single-center study in STEMI patients undergoing primary PCI patients held in Moewardi General Hospital, Central Java, Indonesia. The investigator divided 70 patients with STEMI into two groups, the first is the NAC group, which will get 480 mg of intracoronary NAC immediately after the lesion is opened during primary PCI is performed and the second group will have a normal saline bolus. Each patient will be checked for malondialdehyde, IL-6, hs-troponin I, and caspase-3 just before the primary PCI is performed and 24 hours after intervention. GLS examinations were carried out at admission, discharge, and 6 months after the intervention. The 6MWT examinations were conducted at 1 week and 6 months after the intervention. Furthermore, researchers recorded data on all-cause mortality, rehospitalization, and ACS recurrence at day 30 and 6 months. The study was approved by the hospital ethics committee. The clinical parameters above will then be analyzed. To determine the mean difference between each group (intervention and control) before and after treatment a paired T-test is used if the data distribution is normal (if not, the Wilcoxon test is used). To determine the mean difference between unpaired groups (treatment and control), an independent T-test is used if the distribution is normal (if not, the Mann-Whitney test is used). Normality testing is performed using the Shapiro-Wilk test, considering the sample size is less than 50 per group.

ELIGIBILITY:
Inclusion Criteria:

1. STEMI patients according to The Fourth Universal Definition of Myocardial Infarction from the European Society of Cardiology, American College of Cardiology, American Heart Association, and World Heart Federation Treated by Primary PCI.
2. Aged 30-60 years
3. Willing to participate in the study and sign informed consent.

Exclusion Criteria:

1. Patients with cardiogenic shock (SBP ≤ 80 mmHg, cold extremities, urine output <0.5 ml/kg/hour) <24 hours before randomization
2. Patients with a history of myocardial infarction
3. Patients with a history of chronic heart failure before the onset of AMI
4. Patients scheduled for coronary artery bypass surgery
5. Patients with chronic renal failure or requiring dialysis
6. Patients with chronic inflammation
7. Patients with malignancy
8. Patients with a history of hyper/hypothyroidism
9. Patients with acute infection
10. Patients with sepsis
11. Patients with acute stroke
12. Patients with pulmonary fibrosis
13. Patients with a history of autoimmune disease
14. Patients with a history of anti-inflammatory / antioxidant supplementation
15. Patients with allergy to N-acetylcysteine
16. Pregnant and lactating patients

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-07 (Actual)

PRIMARY OUTCOMES:
Improvements in Biomolecular Parameters (Oxidative Stress) | 24 hours
  Malondialdehyde (ng/L)
Improvements in Biomolecular Parameters (Inflammation) | 24 hours
  Interleukin-6 (ng/L)
Improvements in Biomolecular Parameters (Necrosis) | 24 hours
  high sensitivity troponin I (ng/L)
Improvements in Biomolecular Parameters (Apoptosis) | 24 hours
  Caspase-3 (ng/L)

SECONDARY OUTCOMES:
Improvements in Echocardiographic Parameters | 1 weeks
  Global Longitudinal Strain (%)
Improvements in Physical Parameters | 1 week
  6 Minutes Walking Test (METs)
All-cause mortality | 30-days and 6 months
Rehospitalization | 30-days and 6 months
Recurrent ACS events | 30-days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Yasa, MD, Principal Investigator — Universitas Sebelas Maret; Trisulo Wasyanto, Prof. DR.dr., Principal Investigator — Universitas Sebelas Maret
Locations (1):
- Dr. Moewardi General Hospital, Surakarta, Central of Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
This study was conducted as part of the final project for doctoral program, there was no sponsorship during this study therefore the IPD cannot be shared

REFERENCES:
- [Background] Liu HW, Han YL, Jin QM, Wang XZ, Ma YY, Wang G, Wang B, Xu K, Li Y, Chen SL. One-year Outcomes in Patients with ST-segment Elevation Myocardial Infarction Caused by Unprotected Left Main Coronary Artery Occlusion Treated by Primary Percutaneous Coronary Intervention. Chin Med J (Engl). 2018 Jun 20;131(12):1412-1419. doi: 10.4103/0366-6999.233948. PMID 29893357
- [Background] Yang C, Deng Z, Li J, Ren Z, Liu F. Meta-analysis of the relationship between interleukin-6 levels and the prognosis and severity of acute coronary syndrome. Clinics (Sao Paulo). 2021 Jul 5;76:e2690. doi: 10.6061/clinics/2021/e2690. eCollection 2021. PMID 34231707
- [Background] Aladag N, Asoglu R, Ozdemir M, Asoglu E, Derin AR, Demir C, Demir H. Oxidants and antioxidants in myocardial infarction (MI): Investigation of ischemia modified albumin, malondialdehyde, superoxide dismutase and catalase in individuals diagnosed with ST elevated myocardial infarction (STEMI) and non-STEMI (NSTEMI). J Med Biochem. 2021 Jun 5;40(3):286-294. doi: 10.5937/jomb0-28879. PMID 34177373
- [Background] Rathod KS, Hamshere S, Khambata RS, Andiapen M, Westwood M, Mathur A, Ahluwalia A, Jones DA. Combined analysis of the safety of intra-coronary drug delivery during primary percutaneous coronary intervention for acute myocardial infarction: A study of three clinical trials. JRSM Cardiovasc Dis. 2017 Aug 16;6:2048004017725988. doi: 10.1177/2048004017725988. eCollection 2017 Jan-Dec. PMID 29104752
- [Background] Pasupathy S, Tavella R, Grover S, Raman B, Procter NEK, Du YT, Mahadavan G, Stafford I, Heresztyn T, Holmes A, Zeitz C, Arstall M, Selvanayagam J, Horowitz JD, Beltrame JF. Early Use of N-acetylcysteine With Nitrate Therapy in Patients Undergoing Primary Percutaneous Coronary Intervention for ST-Segment-Elevation Myocardial Infarction Reduces Myocardial Infarct Size (the NACIAM Trial [N-acetylcysteine in Acute Myocardial Infarction]). Circulation. 2017 Sep 5;136(10):894-903. doi: 10.1161/CIRCULATIONAHA.117.027575. Epub 2017 Jun 20. PMID 28634219
- [Background] Hausenloy DJ, Yellon DM. Myocardial ischemia-reperfusion injury: a neglected therapeutic target. J Clin Invest. 2013 Jan;123(1):92-100. doi: 10.1172/JCI62874. Epub 2013 Jan 2. PMID 23281415
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654